CLINICAL TRIAL: NCT01507922
Title: Comparative Efficacy and Safety of Fenoverine and Trimebutine Maleate in Irritable Bowel Syndrome; A Randomized Double-blind Parallel Multi-center Phase IV Trial
Brief Title: Comparative Efficacy and Safety of Fenoverine
Acronym: FEN-401
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FEN-401
Record Dates: First submitted 2012-01-05; First posted 2012-01-11 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Fenoverine; Irritable Bowel Syndrome; Abdominal pain; BSS
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — fenoverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenoverine (Experimental): Fenoverine 100mg three times a day will be administered for 8 weeks.
  Interventions: Drug: Fenoverine
- Trimebutine (Active Comparator): Trimebutine maleate 150mg three times a day will be administered for 8 weeks.
  Interventions: Drug: Timebutine

INTERVENTIONS:
Drug: Fenoverine — Fenoverine 100mg three times a day for 8 weeks
  Other Names: Fexadin
  Arms: Fenoverine
Drug: Timebutine — Timebutine maleate 150mg three times a day for 8 weeks
  Other Names: Polybutin
  Arms: Trimebutine

SUMMARY:
It is a randomized double-blind parallel phase IV study to compare Fenoverine and Trimebutine maleate in the efficacy and safety.

Study Hypothesis: Fenoverine is non-inferior to Trimebutine maleate in its efficacy and safety.

DETAILED DESCRIPTION:
For subjects with IBS, Fenoverine and Trimebutine will be administered orally for 8 weeks; Fenoverine 100mg capsule three times a day and Trimebutine 150mg tablet three times a day. Because one is capsule and the other is tablet, double dummy design will be used. Efficacy is evaluated at the end of 8 weeks and safety will be followed for 4 more weeks after the end of the scheduled medication.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and 60 years of age or younger
* Diagnosed as irritable bowel syndrome using Rome III Criteria
* Female subjects of child-bearing potential are confirmed to have a negative urine beta-hCG test within 7 days prior to administration of initial dose of investigational products.
* Female subjects of child-bearing potential must agree to use contraceptive measures during study period.

Exclusion Criteria:

* Known allergy or hypersensitivity to investigational products or components of the formulation
* Past or current diagnosis of chronic liver disease (e.g., liver cirrhosis, acute hepatitis, alcoholic hepatitis, chronic alcohol abuse and HCC)
* Past or current diagnosis of Myopathy
* Subject with serious renal disease
* Known medical condition assessed by investigators as inappropriate for the study
* Continuous use of NSAIDS, analgesics, steroids, or other immunosuppressants.
* Continuous use of HMG-CoA reductase inhibitors or fibrates to lower blood lipid level
* Pregnant, lactating, or planning to be pregnant women
* Evidence of abuse of drugs or alcohol within 6 months prior to screening
* Participation in other clinical trials within 3 months prior to enrollment or elapse of less than 5 half lives of previous investigational product after last dose of it.
* Unable to submit informed consent or comply with the requirements of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
the proportion of subjects with improvement in abdominal pain or discomfort | week 8
  the proportion of subjects who experienced more than 30% improvement in abdominal pain or discomfort score with visual analog scale at week 8 compared to baseline

SECONDARY OUTCOMES:
BSS scores (each and total) | week 4, 8
  BSS score will be checked for four IBS symptoms; abdominal pain or discomfort, bloating, constipation, diarrhea. The scores will be compared for its chronological changes between trial groups. Total BSS score will be the sum of the scores of four symptoms measured.
overall BSS score | Week 4, 8
  IBS symptom will be assessed overally by subjects at day 1, week 4, and week 8. The scores will be compared chronologically between groups.
subject's satisfaction with treatment | week 4, 8
  Subject's satisfaction with the treatment is measured using visual analog scale.
adverse event | at each visit or contact until 4 weeks after the last dose
  Vital signs will be checked at each visit. Laboratory tests will be conducted at baseline and week 8, and at any time if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Tae Jeen, Dr., Principal Investigator — Korea University Anam Hospital
Locations (7):
- South Korea (7):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Kangwon National University Hospital, Chuncheon
  - Gachon University Gil Hospital, Incheon
  - Inje University Seoul Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul